CLINICAL TRIAL: NCT05053438
Title: Evaluating Hunger Manipulation as an Adjunct to Behavioral Intervention During Intensive Multidisciplinary Feeding Intervention
Brief Title: Evaluating Hunger Manipulation During Feeding Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Valerie M. Volkert, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002492
Record Dates: First submitted 2021-09-01; First posted 2021-09-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Feeding Disorders; Feeding and Eating Disorders; Avoidant/Restrictive Food Intake Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Avoidant Restrictive Food Intake Disorder | interventions — Standard of Care; Nutritional Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to intensive feeding intervention (standard care) or intensive feeding intervention (standard care) + rapid tube weaning study groups using permuted blocks of size 2 or 4.
Who Masked: Investigator
Masking Description: The allocation pattern is concealed to the investigators and therapists providing intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Multidisciplinary Intervention (Standard Care) (Active Comparator): Children with a history of chronic food refusal will be randomized to receive the standard of care. The standard of care for tube wean is to accomplish the balance between enteral supplementation and oral intake, the tube feeding regimen will follow the schedule of therapeutic meals (e.g., mid-day supplementation occurs after morning therapeutic meals).
  Interventions: Behavioral: Intensive Multidisciplinary Feeding Intervention (IMFI)-Standard of Care
- Intensive Multidisciplinary Intervention (Standard Care) + Hunger provocation (Rapid Tube Wean) (Experimental): Children with a history of chronic food refusal will be randomized to receive the experimental arm that combines standard care with rapid tube wean.
  All schedules and documents will be updated accordingly. After the 50% tube wean cut, the dietitian will use regular tube wean sheet to provide credit for oral intake for remainder of admission.
  Interventions: Behavioral: Intensive Multidisciplinary Feeding Intervention (IMFI) standard of care + rapid tube weaning

INTERVENTIONS:
Behavioral: Intensive Multidisciplinary Feeding Intervention (IMFI)-Standard of Care — Standard care involves behavioral intervention delivered during admission Intensive Multidisciplinary Intervention. Patients admitted to the program will participate in four therapeutic meals per day, five days per week (Monday through Friday). The behavioral intervention involves a standard sequence of reinforcement techniques, bite persistence (a.k.a., contingency contacting, escape extinction), and stimulus fading/antecedent manipulation protocols. Parent training will be the central method for structuring meals and transferring treatment gains from the clinic to the home setting. The sequence and steps for parents training will follow a sequential, proficiency-based process, with caregivers transitioning to serve as the primary feeder by discharge.
  Management of tube wean in our standard of care involves reducing tube feeding calories based on oral intake at a 1:1 ratio.
  Other Names: Standard of Care; Nutrition
  Arms: Intensive Multidisciplinary Intervention (Standard Care)
Behavioral: Intensive Multidisciplinary Feeding Intervention (IMFI) standard of care + rapid tube weaning — The experimental arm combines standard care with a rapid tube wean. On day 1, the dietitian will meet with the caregiver to determine the usual tube feeding schedule. The dietitian will then create a tube feeding plan that meets 70% of the child's caloric needs (a 30% reduction).On day 3, if a patient has moved past a rice size bite volume in therapeutic meals, the patient's tube feedings will be further reduced to meet 50% of needs. All schedules and documents will be updated accordingly. After the 50% tube wean cut, the dietitian will use a regular tube wean sheet to provide credit for oral intake for the remainder of admission.
  Other Names: Intervention Group; Rapid Tube Weaning
  Arms: Intensive Multidisciplinary Intervention (Standard Care) + Hunger provocation (Rapid Tube Wean)

SUMMARY:
The primary objective of this study is to determine to what extent hunger provocation, via rapid weaning from enteral feedings, is acceptable and feasible and to evaluate the effect of this intervention when used in an intensive multidisciplinary feeding intervention (IMFI) model of treatment (standard care), for individuals with Avoidant Food Intake Disorder (ARFID) who are dependent on enteral feedings to meet their daily caloric needs.

DETAILED DESCRIPTION:
The recognized standard of care for children dependent on feeding tubes is intensive multidisciplinary feeding intervention (IMFI) involving a professional team that includes psychologists, physicians, nurse practitioners, registered dietitian nutritionists, and speech-language pathologists/occupational therapists working together in inpatient or day hospital settings. A meta-analysis of 11 studies involving intensive, multidisciplinary intervention reported that 71% (95% CI, 54%-83%) of 454 patients successfully weaned from feeding tube dependence at discharge from inpatient or intensive day treatment programs. Treatment gains were maintained following discharge, with 80% (95% CI, 66%-89%) of 414 patients successfully weaned from tube feedings at last follow-up. The most common treatment approaches documented by the meta-analysis involved behavioral intervention and tube weaning (hunger manipulation - evoking a state of hunger to encourage oral consumption by rapidly weaning from the tube). The review highlighted the lack of consensus among clinicians and researchers regarding the criteria for, rate of, and timing of weaning from enteral feedings.

As a result, the authors concluded that the relative contribution of aggressive tube weaning as a standalone or adjunctive therapy to behavioral intervention remains uncertain.

The primary objective of this study is to determine to what extent hunger provocation, via rapid weaning from enteral feedings, is acceptable and feasible and to evaluate the effect of this intervention when used as an adjunct to our standard model of behavioral intervention within the study team's IMFI program, for individuals with Avoidant Food Intake Disorder (ARFID) who are dependent on enteral feedings to meet their daily caloric needs.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 months and 6 years of age;
* Present with dependence on enteral feeding for at least 80% of their daily caloric needs; - Have some prior experience consuming food orally;
* Demonstrate safe and functional swallowing;
* Present without neuromuscular conditions who are non-ambulatory (such as cerebral palsy);
* Have a body mass index in the 15th percentile, or greater;
* Present with no evidence of moderate or severe malnutrition (weight for age or BMI of age z-score < -1) or recent weight loss;
* Engage in no severe problem behavior outside of mealtimes;
* Have a stable sleep schedule that will not interfere with therapeutic meals throughout the day;
* Caregivers must be English-speaking;
* Caregivers must be present for and participate in all treatment sessions.

Exclusion Criteria:

* Individuals with significant active medical conditions requiring oversight from a physician;
* Subjects who display severe problematic behaviors outside of the mealtime, necessitating intervention to specifically address those behaviors; -
* Subjects with medical, structural, or functional limitations preventing safe oral intake of pureed foods;
* Subjects with documented evidence of moderate to severe malnutrition or recent weight loss;
* Individuals with avoidance/restrictive food intake disorders who are not dependent on enteral feedings for at least 80% of their daily caloric needs.

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of oral intake | Up to 12 months
  The percent oral intake will be calculated by dividing calories consumed during therapeutic meals by the daily calorie target.
Percent of patients achieving full wean and time to full wean | Measured in days with a time frame of up to 12 months
  % of participants reaching 100% of their caloric needs by mouth

SECONDARY OUTCOMES:
Change in weight and BMI | Up to 12 months
  Weight will be measured in kilograms (Kg) on a digital scale; height measured in cm; BMI calculated from weight and height into kg/m2, z-score, and percentile
Mealtime performance. | Up to 12 months
  Bite acceptance, rapid swallowing, and inappropriate mealtime behavior

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Volket, PhD, BCBA-D, Principal Investigator — Emory -Children's Ped Institute
Locations (2):
- United States (2):
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - Marcus Autism Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Access to deidentified research data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately after publication.
Access Criteria: The researchers will share the data with anyone who wishes to access the data for any purpose.
  Proposals should be addressed to Dr. Volkert. To gain access, data requestors will need to sign a data access agreement. Data will available for 5 years.